CLINICAL TRIAL: NCT03742193
Title: A Phase II Study of Gemcitabine-docetaxel Chemotherapy With Anti-angiogenic Therapy for Pulmonary Resectable Metastases of Osteosarcoma
Brief Title: Pulmonary Resectable Metastases of Osteosarcoma With Anti-angiogenics and CHemotherapy
Acronym: PROACH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Weibin Zhang, MD, PhD., Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018LLS-NO.84-3
Record Dates: First submitted 2018-09-25; First posted 2018-11-15 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Osteosarcoma; Pulmonary Metastases; Apatinib
MeSH Terms: conditions — Osteosarcoma | interventions — apatinib; Drug Therapy

STUDY DESIGN:
Masking Description: An Independent radiologic reviewing committee assess the radiological tumor response in a blinded manner. Data Safety and Monitoring Board (DSMB) access the outcome in the interim analysis and final analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib + GD group (Experimental): Apatinib + GD regimen. For unilateral metastases,3 cycles before metastasectomy, and 4 cycles after. For bilateral metastases, 3 cycles before first metastasectomy, 1 cycle inbetween, and then second metastasectomy followed by 4 cycles. Apatinib monotherapy is then maintained until 1 year following complete resection.
  Interventions: Drug: Apatinib; Drug: GD regimen

INTERVENTIONS:
Drug: Apatinib — Apatinib 250mg tablet by mouth, bid. 48 hrs break before and 96 hrs after the surgical resection of the pulmonary metastases.
  Other Names: VEGFR Inhibitor
Drug: GD regimen — One cycle: gemcitabine 900 mg/m^2 over 90 min on Day 1, and gemcitabine 900 mg/m^2 and docetaxel 75 mg/m^2 on Day 8. Every 21 days were eligible.
  1~2 -week break before and 2-week break after the surgical resection of the pulmonary metastases is taken.
  Other Names: Chemotherapy

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of Second-line chemotherapy combined with Apatinib for the patients with resectable pulmonary metastasis of osteosarcoma.

DETAILED DESCRIPTION:
After standard chemotherapy and surgery for the localized disease, pulmonary metastases of osteosarcoma occurs in up to 40% of cases and still remain challenging without satisfactory regimen. Apatinib is a oral kinase inhibitor of receptor tyrosine targeting VEGFR2. A pilot study indicated that Apatinib improved the PFS after multi-line chemotherapy failure, and might partly reversed chemo-refractory status for advanced osteosarcoma. Thus, the investigators explored the efficacy of combining Apatinib with current available second-line chemotherapy compared to chemotherapy alone for treating first resectable pulmonary metastases of osteosarcoma following the failure of first-line chemotherapy and wide/radical-margin surgery. Participants will receive 250 mg of apatinib twice daily combined with gemcitabine-docetaxel (GD) regimen before and after the surgical resection of the pulmonary metastases. Osteosarcoma patients with pulmonary recurrence only at baseline will be recruited in the study. The primary end point is progression-free survival rate (PFR) compared with historical control. A12 month PFR of 30% or less is considered inactive, while a 12 month PFR of 50% or greater is regarded as of interest for additional development. With a type I error rate of 5% and a power of 83%, the number of patients needed for this design is 43.

ELIGIBILITY:
Inclusion Criteria:

* age between 10 and 50 years;
* diagnosis of histologically confirmed high grade osteosarcoma;
* identification of pulmonary metastases without the existence of local recurrence(previous re-resection of local recurrence with wide margin is allowed).
* resectable pulmonary nodule(s), defined as nodule(s) that are removable by wedge resection/ segmentectomy/lobectomy without necessitating a pneumonectomy (e.g., nodules immediately adjacent to the main stem bronchus or main pulmonary vessels)
* prior treatment consisted of standard National Comprehensive Cancer Network (NCCN) guideline recommended first-line chemotherapy
* wide/radical-margin surgical resection of the primary tumor completed at least 4 weeks before enrollment.
* Eastern Cooperative Oncology Group(ECOG) performance status 0-2 with a life expectancy >3 months;
* adequate renal, hepatic, and hemopoietic function;
* normal or controlled blood pressure;
* no thoracic comorbidities with adequate pulmonary function eligible for thoracic surgery

Exclusion Criteria:

* previously exposed to GD chemotherapy or VEGFR2 Tyrosine-kinase inhibitors (TKIs);
* existence of local recurrence;
* have had other kinds of malignant tumors at the same time;
* cardiac insufficiency or arrhythmia;
* uncontrolled complications, such as diabetes mellitus and so on;
* coagulation disorders or Hemorrhagic diseases ;
* metastases considered unresectable or borderline resectable at baseline
* intolerable of thoracis surgery
* pleural or peritoneal effusion that needs to be handled by surgical treatment;
* combined with other infections or wounds
* wound dystrophy, poor soft-tissue around implantation or other wound complications risky of non-healing given angiogenesis inhibitor assessed by the investigators

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Estimated)
Dates: Start 2019-08-11 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
12 months Progression-free survival rate(12mPFR) | 12 months from the recruitment of the study
  The proportion of patients with progression-free survival at 12 months according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1). A 12mPFR of 30% or less is considered inactive, while a 12mPFR of 50% or greater is regarded as of interest for additional development

SECONDARY OUTCOMES:
Overall survival (OS) | Baseline until death, followed through study completion, an average of 2 years
  calculated from the date of treatment start until last follow-up or death, whichever comes first.
Total resectability | after neoadjuvant systemic therapy, an average of 8~9 weeks
  The number of patients undergoing pre-planned metastasectomy divided by the number of patients considered resectable at baseline
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion, an average of 1 years
  The occurrence of each adverse events(AEs), severe AEs(SAEs) and death according the CTCAE_5.0
Objective response rate (ORR) | after neoadjuvant systemic therapy, an average of 8~9 weeks
  Complete Response(CR)+Partial Response(PR) after neoadjuvant systemic therapy
Clinical benefit rate (CBR) | after neoadjuvant systemic therapy, an average of 8~9 weeks
  CR+PR+stable disease (SD) after neoadjuvant systemic therapy
Progression free survival (PFS) | Baseline until disease progression or death, whichever occurs first (followed through study completion, an average of 1.5 years)
  Progression free survival according to RECIST 1.1
OS rate | 12 and 24 months from baseline
  the proportion of OS at 12, 24 months

OTHER OUTCOMES:
Exploratory outcome: Subgroup analysis of progression-free survival(PFS) | Baseline until disease progression or death, whichever occurs first (followed through study completion, an average of 1.5 years)
  The PFS for each subgroups in terms of clinicopathological characteristics (age, gender, histological type, solitary or multiple metastases, unilateral or bilateral metastases, early or late metastases, calcifying or non-calcifying lesions, with or without lesion cavitation, with or without AEs [especially pneumothorax, hand-foot skin reactions, hair depigmentation], etc)
Exploratory outcome: The correlation of potential pathological biomarker with PFS | Baseline until disease progression or death, whichever occurs first (followed through study completion, an average of 1.5 years)
  The correlation between the expression of VEGFR2, CD34, Ki-67 and immune cell infiltration by immunohistochemistry and PFS
Exploratory outcome: Tumor response pre-metastasectomy as a predictor of PFS | Baseline until disease progression or death, whichever occurs first (followed through study completion, an average of 1.5 years)
  to compare the PFS of the three group according to tumor response pre-metastasectomy (group1: CR/PR, group2: SD, group3 PD)
Exploratory outcome: Tumor cavitation as a prognostic factor for oncological outcome | Baseline until disease progression or death, whichever occurs first (followed through study completion, an average of 1.5 years)
  to compare the predictive value of the Crabb's modified RECIST criteria with the original RECIST 1.1 criteria in terms of PFS and OS
Exploratory outcome: AEs of the targeted therapy as prognostic factors for oncological outcome, especially pulmonary lesion cavitation/pneumothorax and hair depigmentation | Baseline until disease progression or death, whichever occurs first (followed through study completion, an average of 1.5 years)
  to correlate the incidence of targeted therapy related AEs （especially pneumothorax, hand foot skin reactions, skin and hair depigmentation and fatigue）with the PFS/OS for the treatment arm.
Correlation of KDR 604 polymorphism with pulmonary lesion cavitation/pneumothorax and with PFS | Baseline until disease progression or death, whichever occurs first (followed through study completion, an average of 1.5 years)
  According to our previous retrospective analysis, we aim the validate the correlation of KDR 604 AA，AG，GG genotype with the incidence of pulmonary lesion cavitation/pneumothorax and PFS among all patients.
Exploratory outcome: 1.0-mm CT scan for the early identification small lung nodule as pulmonary recurrence | Baseline until disease progression or death, whichever occurs first (followed through study completion, an average of 1.5 years)
  to compare the diagnostic value of the 1.0 mm versus 5.0 mm CT scan for the radiological evaluation of small lung nodule as tumor recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Weibin Zhang, PhD, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data of IPD is available to researcher's upon reasonable request, in accordance to the local legislator's policy ( such as genetic sequencing data)